CLINICAL TRIAL: NCT04193930
Title: Soft Versus Conventional Protocol in Ovarian Stimulation in Intracytoplasmic Sperm Injection Cycles for Poor Responders
Brief Title: Different Protocols in Ovarian Stimulation in Intracytoplasmic Sperm Injection Cycles
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: no women were recruited
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohammed Khairy Ali, Lecturer, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ICSI_PR
Record Dates: First submitted 2019-12-07; First posted 2019-12-10 (Actual); Last update posted 2022-11-30 (Actual); Status verified 2022-11

CONDITIONS: ART
MeSH Terms: interventions — Letrozole; Menotropins

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Soft ovarian stimulation protocol (Other)
  Interventions: Drug: Letrozole; Drug: Menotropins
- conventional ovarian stimulation protocol (Other)
  Interventions: Drug: Menotropins; Drug: recombinant Follicular stimulating hormone

INTERVENTIONS:
Drug: Letrozole — Oral tablet letrozole 2,5 mg/twice daily for 5 days
  Arms: Soft ovarian stimulation protocol
Drug: Menotropins — 150 IU of highly purified menotropins intramuscular
Drug: recombinant Follicular stimulating hormone — recombinant Follicular stimulating hormone 300- 400 IU
  Arms: conventional ovarian stimulation protocol

SUMMARY:
During assisted reproduction technology treatments like in vitro fertilization, some patients give a poor ovarian response to controlled ovarian hyperstimulation. The European Society of Human Reproduction and Embryology consensus defined poor response to ovarian stimulation during in vitro fertilization with Bologna criteria.

Bologna criteria: At least two of the following three features must be present:

(i) Advanced maternal age (≥40 years). (ii) Previous Poor responders (≤3 oocytes with a conventional stimulation protocol).

(iii) An abnormal ovarian reserve test Most controlled ovarian hyperstimulation regimens currently used for expected poor responders are based on using a high daily dose (300- 450 IU/day) of exogenous gonadotropins. Giving a high gonadotropin dose obviously increases the cost of in vitro fertilization, a consequence that would be acceptable if paralleled by an improvement in in vitro fertilization outcome. Unfortunately, however, the available data suggest that increasing the daily gonadotropins dose may increase the number of retrieved oocytes, but not the final success rate of in vitro fertilization.

ELIGIBILITY:
Inclusion Criteria:

* Advanced maternal age (≥40 years) .
* Previous Poor responders (≤3 oocytes with a conventional stimulation protocol).
* An abnormal ovarian reserve tests

Exclusion Criteria:

* Hyper or Normal responders patients.
* Endocrine or metabolic diseases like hyperprolactinoma, hypothyroidism,...etc
* Patients with a severe male factor abnormality. 4-Patients with systemic disease such as chronic renal disease, chronic liver disease, etc

Ages: 40 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-01-01 (Actual); Study Completion 2021-01-01 (Actual)

PRIMARY OUTCOMES:
Total gonadotrophins dose | 14 days

SECONDARY OUTCOMES:
Duration of ovarian stimulation | 14 days
Endometrial thickness | 14 days
  by ultrasounds

CONTACTS AND LOCATIONS:
Locations (1):
- Women Health Hospital - Assiut university, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided